CLINICAL TRIAL: NCT04552574
Title: A Clinical Trial to Identify the Effects of HMR(Home Meal Replacement)-Type Medifood on Chronic Metabolic Disorders Including Lipid Metabolism Disorders and Sarcopenia
Brief Title: Randomized Clinical Trial of HMR(Home Meal Replacement)-Type Omega-3-balanced-diet
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chungbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Yonghwan Kim, Clinical Assistant Professor, Chungbuk National University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CBNUH202006021
Record Dates: First submitted 2020-09-13; First posted 2020-09-17 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Chronic Metabolic Disorder; Lipid Metabolism Disorders; Sarcopenia
MeSH Terms: conditions — Lipid Metabolism Disorders; Sarcopenia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): All subjects will intake HMR(Home meal replacement)-type omega-3-balanced-diet for 4 weeks.
  Interventions: Dietary Supplement: HMR(Home meal replacement)-type omega-3-balanced diet
- Control group (No Intervention): No intervention for 4 weeks.

INTERVENTIONS:
Dietary Supplement: HMR(Home meal replacement)-type omega-3-balanced diet — A diet of which omega-3 to omega-6 ratio is below 1:4 was developed by Agricultural entity Green Grass Co., Ltd.. A committee of experts that is composed of several university professors in authorities of IPET(Institute of Planning and Evaluation for Technology in food, agriculture and forestry) also participated in the development of this diet.
  Arms: Intervention group

SUMMARY:
Investigate whether HMR(Home meal replacement)-type omega-3-balanced-diet can improve clinical laboratory values related to chronic metabolic diseases through reducing lipids and chronic inflammation, and can prevent muscle loss.

DETAILED DESCRIPTION:
Korea is entering an post-aged society with an increase in single-person households, and as the average life expectancy increases, the increase in the population exposed to chronic metabolic diseases requires basic dietary solutions for life seeking physical, mental and social well-being. As a result of a survey conducted by the Korean Health Insurance Corporation (2010), medical expenses for chronic metabolic diseases were estimated at 15,233.8 billion won, with 54.3% of adults with chronic diseases, 68.7% in their 50s, 83.7% in their 60s, and 91.3% in their 70s or older. This trend continues to increase, resulting in an increasing social burden. Our researchers focused on functional lipids which provide specific health benefits when ingested to prevent these chronic diseases. Omega 3 is an essential fatty acid that can not be synthesized in the body, maintaining the structure of cells in the human body, helping smooth metabolism. It also inhibits the aggregation of platelets and lowers the risk of coronary artery or cardiovascular disease by lowering the level of neutrality, it has been reported to have an inflammatory mitigation effect. Omega 6 has been reported to cause increased inflammation and ulticaria, asthma, cardiovascular disease side effects when intake is increased. In this context, the recommended ratio of omega 3 and omega 6 is reported to be within 1:4.

A diet of which omega-3 to omega-6 ratio is below 1:4 was developed by Agricultural entity Green Grass Co., Ltd. for prevention of sarcopenia and chronic metabolic disease.

Subjects assigned to the test group receive a total of 4 weeks HMR medifood and consume a regular diet for the next four weeks after having a wash-out period for a total of two weeks. On the other hand, subjects assigned to the control group would be able to consume a regular diet for the first four weeks and take HMR medifood for the next four weeks after having a two-week wash-out period.

ELIGIBILITY:
Inclusion Criteria:

* BMI(Body mass index): 25-40 kg/m2
* Circumference of waist: ≥90 cm in men and ≥85 cm in women
* sBP(systolic Blood pressure): 100-180mmHg
* dBP(diastolic Blood pressure): 70-110mmHg
* Alcohol consumption: ≤14 glasses/week in men and ≤7 glasses in women

Exclusion Criteria:

* Ongoing administration of antihypertensive drugs
* Past medical history of diabetes, dyslipidemia, cardiocerebrovascular disease, or ongoing administration of drugs related to the aforementioned diseases
* Allergies to dairy products or other foods
* Smokers
* Subjects who intend to lose weight in-between during the period of clinical trial
* Abnormal at the screening blood test(AST(Aspartate transaminase), ALT(Alanine transaminase)>100 IU/L, TG(triglyceride)>400 mg/dL, total cholesterol>300 mg/dL, LDL(Low-density lipoprotein)-cholesterol>190 mg, WBC>10000/μL or <1500/μL, hsCRP>5 mg/L)
* Pregnant or breastfeeding women

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2020-08-19 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Lipids | 4 weeks
  LDL(Low-density lipoprotein)-cholesterol and HDL(High-density lipoprotein)-cholesterol
triglyceride | 4 weeks
  Lipids
Muscle mass | 4 weeks
  SLM (Soft lean mass)

SECONDARY OUTCOMES:
WBC (White blood cell) count | 4 weeks
  Inflammation
hsCRP (high-sensitivity C-reactive protein) | 4 weeks
  Inflammation
Balance between omega-3 fatty acids and omega-6 fatty acids | 4 weeks
  Omega-3 fatty acids to omega-6 fatty acids ratio

CONTACTS AND LOCATIONS:
Overall Officials: Jae Hyun Ahn, Study Director — Chungbuk National University Hospital
Locations (1):
- Chungbuk National University Hospital, Cheongju-si, North Chungcheong, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee JW, Kim Y, Hyun T, Song S, Yang W, Kim YS, You HS, Chang YC, Shin SH, Kang HT. Beneficial Effects of a Specially Designed Home Meal Replacement on Cardiometabolic Parameters in Individuals with Obesity: Preliminary Results of a Randomized Controlled Clinical Trial. Nutrients. 2021 Jun 24;13(7):2171. doi: 10.3390/nu13072171. PMID 34202690